CLINICAL TRIAL: NCT04182581
Title: A Study of B-cell Maturation Antigen/Cluster of Differentiation Antigen 19 Dual-Target Chimeric Antigen Receptor T Cell Immunotherapy for Relapsed or Refractory Multiple Myeloma
Brief Title: A Study of BCMA/CD19 Dual-Target CAR-T Cell Immunotherapy for Relapsed or Refractory Multiple Myeloma
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xijing Hospital (Other)
Collaborators: Gracell Biotechnology Ltd. (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PGC0008
Record Dates: First submitted 2019-11-27; First posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-10

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR-T treatment group (Experimental): The patients will receive one dose of BCMA/CD19 dual-target CAR-T. BCMA/CD19 dual-target CAR-T dosage ranges from 5×10^4 to 3×10^5 CAR+T/Kg.
  Interventions: Biological: BCMA/CD19 Dual-Target CAR-T

INTERVENTIONS:
Biological: BCMA/CD19 Dual-Target CAR-T — BCMA/CD19 Dual-Target CAR-T target both BCMA and CD19. The subjects will receive CAR-T as one dose. The dosage ranges from 5×10^4 to 3×10^5 CAR+T/Kg.

SUMMARY:
The study is an early, open, single-centered trial. The purpose of this study is to evaluate the safety and persistence of BCMA/CD19 dual-target CAR-T cell immunotherapy in relapsed or refractory MM. The study will include 18 subjects to receive BCMA/CD19 dual-target CAR-T therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-70 years;
2. Diagnosis of relapsed or refractory multiple myeloma(MM): 1) measurable disease at screening as defined by any of the following: serum monoclonal paraprotein (M-protein) level ≥1.0 g/dL or urine M-protein level ≥200 mg/24 hours; or light chain MM without measurable disease in the serum or the urine: serum immunoglobulin free light chain ≥10 mg/dL and abnormal serum immunoglobulin kappa/lambda free light chain ratio. Light chain MM without measurable disease in the serum or the urine is a specific definition in this study, which refers to subjects whose M-protein in the serum and M-protein in the urine is undetectable; 2) received at least 2 standard regimens, determined as progressive disease (PD) by IMWG criteria; received at least 3 prior lines of treatment for MM, undergone at least 1 complete cycle of treatment for each line, unless PD was documented by IMWG criteria as the best response to the regimen; 3) received a proteasome inhibitor(PI) and an immunomodulatory therapy (IMiD); 4) documented disease progression during, or within 12 months of, most recent anti-myeloma therapy.
3. Histologically confirmed positive expression of CD19 and/or BCMA 3 months prior to enrollment;
4. Eastern cooperative oncology group (ECOG) performance status of 0 to 1;
5. Adequate organ function is defined as: 1) hemoglobin≥8.0g/dL(did not receive red blood cell transfusion ≤7 days prior to laboratory tests; recombinant human erythropoietin is allowed); 2) platelet count >50×10^9/L(did not receive blood transfusion ≤7 days prior to laboratory tests); 3) ANC ≥0.75×10^9/L(did not receive supportive treatment ≤7 days prior to laboratory tests; growth factors are allowed); 4) total bilirubin <2×ULN (for subjects with congenital hyperbilirubinemia such as Gilbert's syndrome, direct bilirubin≤1.5×ULN); 5) creatinine clearance (according to MDRD formulas or 24h urine collection result) ≥40 mL/min/1.73m^2; 6) ALT and AST <3×ULN; 7) corrected serum calcium ≤12.5 mg/dL (≤3.1 mmol/L), or free calcium ion ≤6.5 mg/dL(≤1.6 mmol/L); 8) oxygen saturation >92% on non-oxygen-assistance state;
6. Females of childbearing potential must have a negative serum hypersensitive β-human chorionic gonadotropin (β-hCG) or urine pregnancy test result, at screening, and prior to lymphodepletion;
7. Females of childbearing potential must agree to use a highly effective contraception continuously from signing informed consent form until ≥100 days after CAR-T infusion (when continuously correctly used, failure rate <1% per year). Highly effective contraception include, user-independent method: 1) implantable progesterone contraceptives which can inhibit ovulation; 2) intrauterine device (IUD); Intrauterine hormone release system; 3) partner has a vasectomy; user-dependent method: 1) compound hormone contraceptives which can inhibit ovulation (contain estrogen and progesterone, oral/vaginal/transdermal administration); 2) progesterone contraceptives which can inhibit ovulation (oral administration or injection);
8. Except for highly effective contraception, males must agree to use barrier contraception (such as condom plus spermicidal foam/gel/film/suppository) during sexual contact with a female of childbearing potential, to use condom during sexual contact with a pregnant female, from signing informed consent form until ≥100 days after CAR-T infusion; females and males must agree to avoid ovum/oocyte/sperm donation, during the study period and ≥100 days after CAR-T infusion. Note: hormone contraceptives may interact with the study treatment, thus reducing the contraceptive effect;
9. Subject must sign an inform consent form indicating that he or she understands the purpose of and procedures required for the study and is willing to participate in the study. Consent is to be obtained prior to the initiation of any study-related tests or procedures that are not part of standard-of-care for the subject's disease;
10. Willing and able to adhere to the prohibitions and restrictions specified in this protocol.

Exclusion Criteria:

1. History of CAR-T treatment, the target of CAR-T is not limited;
2. History of anti-CD19 or anti-BCMA treatment;
3. Concomitant invasive malignancy other than diagnosis or treatment of other radically-cured malignancies without malignant change ≥3 years prior to enrollment or adequately- treated non-melanoma skin cancer without malignant change evidence;
4. Received targeted therapy, epigenetic therapy, experimental drug therapy, or experimental invasive medical device <14 days or 5 half-lives (according to the shorter one) prior to leukapheresis; received monoclonal antibody <21 days prior to leukapheresis; received cytotoxic chemotherapy, PI, radiotherapy <14 days prior to leukapheresis (for radiotherapy, if the radiation field is no more than 5% of bone marrow reserve, whenever radiotherapy ended, the subject is allowed to participate in the study); received IMiD <7 days prior to leukapheresis;
5. Toxicities related to prior therapy did not relieve to baseline or ≤ grade 1, except for peripheral neuropathy and alopecia;
6. The following cardiac conditions: New York Heart Association(NYHA) grade III or IV congestive heart failure; myocardial infarction or coronary artery bypass graft (CABG) ≤6 months prior to enrollment; history of clinically significant ventricular arrhythmia or unexplained syncope, not believed to be vasovagal in nature or due to dehydration; history of severe non-ischemic cardiomyopathy; impaired cardiac function (LVEF <45%) as assessed by echocardiogram or multiple-gated acquisition (MUGA) scan (performed ≤ 8 weeks prior to leukapheresis);
7. Systemic or local corticosteroid therapy of greater than 5 mg/day of prednisone (or equivalent dose of another corticosteroid) within 2 weeks prior to leukapheresis;
8. Received either of the following: an allogeneic stem cell transplant for MM; an autologous stem cell transplant ≤ 12 weeks prior to leukapheresis;
9. Known active central nervous system (CNS) involvement or emergence of meninges involvement clinical signs;
10. Stroke or convulsions ≤ 6 months prior to ICF signing;
11. Presence of plasma cell leukemia(plasma cell >2.0×10^9/L), Waldenstrom's macroglobulinemia, POEMS syndrome(polyneuropathy, organomegaly, endocrinopathy, monoclonal protein disease, skin changes) or primary amyloidosis(AL) at screening;
12. Seropositive for human immunodeficiency virus (HIV); Hepatitis B infection as defined according to the American Society of Clinical Oncology (ASCO) guidelines. In the event the infection status is unclear, quantitative levels are necessary to determine the infection status. Hepatitis C (anti-hepatitis C virus [HCV] antibody positive or HCV-RNA quantitation positive) or known to have a history of hepatitis C;
13. Attenuated live vaccine ≤4 weeks prior to enrollment;
14. Known life threatening allergies, hypersensitivity, or intolerance to CAR-T cells or its ingredients, including dimethylsulfoxide;
15. Serious underlying medical condition, such as: evidence of serious active viral, bacterial, or uncontrolled systemic fungal infection; active autoimmune disease or a history of autoimmune disease within 3 years; overt clinical evidence of dementia or altered mental status; hereditary bleeding/ coagulating disease, a history of non-traumatic bleeding or thromboembolism, other disease that may increase bleeding risk;
16. Presence of any problems that may be detrimental to the subjects' receiving/tolerating planned treatment and the subject's understanding ICF; presence of any condition that the investigators think it is inappropriate for the subject to anticipate the trial (such as damaging health); presence of any condition that may deter, limit, or obfuscate protocol-defined evaluation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-10-15 (Actual); Primary Completion 2020-09 (Estimated); Study Completion 2021-05 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of treatment related AE | 2 years
  Adverse events(AEs) will be collected and graded according to ASTCT consensus(for Cytokine Release Syndrome, CRS and Immune Effector Cell-Associated Neurotoxicity Syndrome, ICANS) and CTCAE v5.0(for AE except CRS/ICANS ).
Incidence of DLT | 12 weeks
  Dose-limiting toxicity (DLT) will be collected. DLT refers to toxicity that limit the process to continue increasing CAR-T dose.
CAR copies concentration in peripheral blood | 2 years
  CAR copies in peripheral blood will be measured by qPCR and FCM.

SECONDARY OUTCOMES:
ORR | 2 years
  Objective response rate (ORR) will be calculated. ORR refers to the proportion between the number of subjects who are evaluated as PR or status better than PR and total number of subjects.
DOR | 2 years
  Duration of response (DOR) will be calculated. DOR refers to the time between the initial response (CR or PR) to therapy and evaluated as PD for the first time or death due to any reason.
PFS Rate | 2 years
  Progression free survival (PFS) rate will be calculated. PFS refers to the proportion between the number of subjects who are evaluated as PD or died and total number of subjects.
OS Rate | 2 years
  Overall survival (OS) rate will be calculated. OS refers to the proportion between the number of subjects who died and total number of subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Xiequn Chen, Doctor, Principal Investigator — First affiliated hospital of air force military medical university(i.e., Xijing Hopital)
Locations (1):
- First affiliated hospital of air force military medical university(i.e., Xijing Hopital), Xi’an, Shanxi, China